CLINICAL TRIAL: NCT06162078
Title: A Baseline Epidemiological Study to Document the Malaria Burden in Pregnant Women and the Incidence of Pregnancy in a Cohort of Nulligravida to Targeted Futur Malaria Vaccine Candidate Efficacy in Pregnancy in Burkina Faso
Brief Title: Malaria Burden in Pregnant Women and the Incidence of Pregnancy in a Cohort of Nulligravida
Acronym: EPI-PAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe de Recherche Action en Sante (Other)
Collaborators: European Vaccine Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: GRAS
Record Dates: First submitted 2023-07-25; First posted 2023-12-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Maternal Malaria During Pregnancy - Baby Not Yet Delivered

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subgroup 1, Household longitudinal survey of nulligravida cohort: fieldworkers will visit the households in the study area to identify and enroll women meeting the eligibility criteria. After consenting a fingerprick blood sample will be obtained for pregnancy testing and malaria blood smear, and VAR2CSA antibodies measurement. Enrolled women will be visited every trimester to check for pregnancy and malaria infection. The follow up of each participant will end upon a pregnancy test is positive or at month 9 after the enrolment.
- Subgroup 2, Single timepoint evaluation for primigravidae 1rst, 2nd and 3 rd trimester: Participants will be enrolled by study staff stationed at the antenatal care clinic. Women attending the ANC visit at any gestational age will be screened and those meeting the eligibility criteria will undergo the study procedures which includes collecting demographic data, medical and pregnancy history. They will then be requested to donate a fingerprick blood sample for malaria infection and hemoglobin measurement.
- Subgroup 3, Single timepoint evaluation at primigravidae delivery: participants will be recruited during any of the ANC visit as consenting process will not be feasible during the labour at delivery. They will be issued a sticker that will be affixed to the health card so that they could easily be recognized when they come for delivery.
  At delivery, samples will be collected from fingerprick, cord blood and placenta for detecting malaria infection by microscopy and histopathology. Additional data will be collected on the neonate for secondary outcomes assessment, adverse birth outcomes .

SUMMARY:
The overarching aims of this study are to longitudinally determine the occurrence of pregnancy in a cohort of nulligravida at the community level and to estimate the burden of malaria infection during the course of the pregnancy till delivery.

DETAILED DESCRIPTION:
Three subgroups will involve in the design of this study:

for subgroup 1, fieldworkers will visit the households in the study area to identify and enroll women meeting the eligibility criteria to involve in a nulligravida cohort aged ≥ 15 years. After consenting a fingerprick blood sample will be obtained for pregnancy testing, malaria blood smear, and VAR2CSA antibodies measurement. Enrolled women will be visited every trimester to check for pregnancy and malaria infection. The follow up of each participant will end upon a pregnancy test is positive or at month 9 after the enrolment.

Participants to subgroup 2 will be enrolled primigravidae aged ≥ 15 years by study staff stationed at the antenatal care clinic. Women attending the ANC visit at any gestational age will be screened and those meeting the eligibility criteria will undergo the study procedures which includes collecting demographic data, medical and pregnancy history. They will then be requested to donate a fingerprick blood sample for malaria infection and hemoglobin measurement. This will be a single timepoint evaluation.

Subgroup 3 participants will be recruited primigravidae aged ≥ 15 years during any of the ANC visit as consenting process will not be feasible during the labour at delivery. They will be issued a sticker that will be affixed to the health card so that they could easily be recognized when they come for delivery. At delivery, samples will be collected from fingerprick, cord blood and placenta for detecting malaria infection by microscopy and histopathology. Additional data will be collected on the neonate for secondary outcomes assessment.

ELIGIBILITY:
Inclusion Criteria:

* For subgroup 1

  * Nulligravidae aged ≥ 15 years
  * Residing within the study area and planning to stay for the study duration
  * Signed or thumb-printed informed consent obtained from participant/participant legally acceptable representatives. An assent will be obtained from minors.
* For subgroups 2 and 3

  * Primigravidae aged ≥ 15 years at the time of enrolment
  * Residing within the study area for the last three months
  * Signed or thumb-printed informed consent obtained from participant/participant legally acceptable representatives. An assent will be obtained from minors.
* Additional criteria for subgroup 3 • Third trimester of gestational age

Exclusion Criteria:

* For subgroup 1 only

  * Women of non-childbearing potential. Non-childbearing potential is defined as current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
  * Women reporting established use of oral, injected or implanted hormonal contraceptives; intrauterine device or intrauterine system
* For all the subgroups

  * Chronic use of i) immunosuppressive drugs, ii) or other immune modifying drugs within three months prior to enrolment in the study
  * Known history of Human Immunodeficiency Virus (HIV) (No test will be done by the study)
  * Use of any other investigational or non-registered product (drug or vaccine) during the study period.
  * Any previous participation in any malaria (vaccine) study.
  * Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female nulligravida able to become pregnant for sub-group 1 and primigravidae attending to ANC or deliver
Study Population: For subgroup 1:
  Fieldworkers will visit the households in the study area to identify and enroll women meeting the eligibility criteria.
  For subgroup 2:
  Paticipants will be enrolled by study staff stationed at the antenatal care clinic. Women attending the ANC visit at any gestational age will be screened and enrolled.
  For Subgroup 3:
  Participants will be recruited during any of the ANC visit as consenting process will not be feasible during the labour at delivery. They will be issued a sticker that will be affixed to the health card so that they could easily be recognized when they come for delivery.
Sampling Method: Probability Sample
Enrollment: 2390 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of nulliparous with positive urine test | 9 months
  Proportion of nulliparous with positive urine pregnancy test at 3 months, 6 months and 9 months post enrolment
P. falciparum infection in nulliparous attending the antenatal care visit | 9 months
  Prevalence of P. falciparum infection by microscopy and PCR (polymerase chain reaction) in nulliparous attending the antenatal care visit at the local health care facility
Moderate and severe anemia during the last antenatal care visit | 9 months
  Proportion of pregnant women with moderate and severe anemia during the last antenatal care visit at the local health care facility
P. falciparum infection at delivery | 9 months
  Prevalence of parasitemia at delivery (maternal and cord blood) by microscopy
Placental infection | 9 months
  Proportion of women at delivery with histopathologically confirmed placental infection

SECONDARY OUTCOMES:
Adverse birth outcomes | 9 months
  Prevalence of adverse birth outcomes (spontaneous abortion, stillbirth, low birth weight (<2,500 g), preterm delivery (<37 weeks))
Uptake IPTp-SP (Intermittent preventive treatment of malaria in pregnancy using sulfadoxine-pyrimethamine) during the pregnancy | 9 months
  Proportion of pregnant women receiving one, two, three and ≥ 3 doses of IPT-SP during the pregnancy

OTHER OUTCOMES:
Titers of VAR2CSA (a large 350-kDa protein comprising six Duffy-binding-like (DBL) domains and three larger interdomain regions) antibodies in nulliparous | 3 months
  Geometric mean titers of VAR2CSA antibodies at enrolment of nulliparous
Gametocytes presence in placental tissue | 9 months
  Gametocytes prevalence in placental tissue
Prevalence of mutations among pregnancy | 9 months
  Prevalence of dhps K540E, dhps A581G and dhfr I164L mutations (Markers of sulfadoxine-pyrimethamine resistance)

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse OUEDRAOGO, MD, PhD, Principal Investigator — Groupe de Recherche Action en Sante (GRAS)
Locations (1):
- GRAS-Banfora, Banfora, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: data available
Access Criteria: publication